CLINICAL TRIAL: NCT02483078
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Trial, Followed by Single-arm Treatment of PRO 140 in Combination With Optimized Background Therapy in Treatment-Experienced HIV-1 Subjects
Brief Title: Randomized, Double-Blind, Placebo-Controlled Trial, Followed by Single-Arm Treatment of PRO 140
Acronym: PRO140
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CytoDyn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO 140_CD 02
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Results first posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: HIV
MeSH Terms: interventions — leronlimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRO 140 (Active Comparator): PRO140 350mg weekly SC Inj. + existing ART for one week. After one week, all subjects will enter the 24-week single-arm, open-label treatment period. During this period, all subjects will receive PRO 140 SC injection and Optimized Background Therapy.
  Interventions: Drug: PRO 140; Drug: Optimized Background Regimen
- Placebo (Placebo Comparator): Placebo weekly SC Inj. + existing ART for one week. After one week, all subjects will enter the 24-week single-arm, open-label treatment period. During this period, all subjects will receive PRO 140 SC injection and Optimized Background Therapy.
  Interventions: Drug: Placebo; Drug: Optimized Background Regimen

INTERVENTIONS:
Drug: PRO 140 — PRO 140 is a humanized IgG4,κ monoclonal antibody (mAb) to the chemokine receptor CCR5.
  Other Names: PRO140, CCR5 antagonist, Humanized monoclonal antibody to CCR5
  Arms: PRO 140
Drug: Placebo
  Arms: Placebo
Drug: Optimized Background Regimen — Optimized background therapy (OBT) is chosen on the basis of a subject's resistance test results and treatment history.
  Other Names: Optimized background therapy (OBT) is chosen on the basis of a subject's resistance test results and treatment history.

SUMMARY:
This is a Phase 2b/3, multi-center, two part study, designed to evaluate the efficacy, safety, and tolerability of PRO 140 in conjunction with existing ART (failing regimen) for one week and Optimized Background Therapy (OBT) for 24 weeks respectively. Study population includes treatment-experienced HIV-infected patients with CCR5-tropic virus who demonstrates evidence of HIV-1 replication despite ongoing antiretroviral therapy with documented genotypic or phenotypic resistance to ART drugs within three drug classes (or within two or more drug classes with limited treatment options).The options may be limited as a result of drug antiviral class cross-resistance or documented treatment intolerance.

DETAILED DESCRIPTION:
PRO 140, in combination with other antiretroviral agents, is indicated for treatment experienced adult HIV-1 patients infected with CCR5-tropic virus. These patients must demonstrate evidence of HIV-1 replication despite ongoing antiretroviral therapy and have documented genotypic or phenotypic resistance to at least one ART drug within three drug classes (or within two or more drug classes with limited treatment option). The options may be limited as a result of drug antiviral class cross-resistance, documented treatment intolerance, documented objective assessments such as renal or hepatic insufficiency (e.g. high creatinine at baseline, limiting treatment options due to potential for toxicity), past adverse reactions such as hypersensitivity reactions or neuropsychiatric issues that could limit use of currently approved drugs.

Study population includes treatment-experienced HIV-infected patients with CCR5-tropic virus who demonstrates evidence of HIV-1 replication despite ongoing antiretroviral therapy with documented genotypic or phenotypic resistance to ART drugs within three drug classes (or within two drug classes with limited treatment option).

Enrollment will be stratified to have HIV-1 virus resistant to ART drugs within three drug classes or within two drug classes with limited treatment option.

The primary objective is to assess the efficacy, clinical safety and tolerability parameters of PRO 140 compared to placebo in reducing HIV-1 viral load during the 1-week double-blind treatment period. The secondary objectives of the trial are to assess the efficacy, clinical safety and tolerability parameters of PRO 140 in combination with Optimized Background Therapy during the 24-week single-arm, open-label treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age ≥ 18 years
2. Exclusive CCR5-tropic virus at Screening Visit
3. Have a history of at least 3 months on current antiretroviral regimen
4. Treatment-experienced HIV-infected patients with documented genotypic or phenotypic resistance to at least one ART drug within three drug classes

   OR

   Treatment-experienced HIV-infected patients with documented genotypic or phenotypic resistance to at least one ART drug within two drug classes and have limited treatment options. The options may be limited as a result of drug antiretroviral class cross-resistance or documented treatment intolerance.
5. Be willing to remain on treatment without any changes or additions to the OBT regimen, except for toxicity management or upon meeting criteria for treatment failure.
6. Plasma HIV-1 RNA ≥ 400 copies/mL at Screening Visit and documented detectable viral load (HIV-1 RNA >50 copies/ml) within the last 3 months prior to Screening Visit.
7. Laboratory values at Screening of:

   * Absolute neutrophil count (ANC) ≥ 750/mm3
   * Hemoglobin (Hb) ≥ 10.5 gm/dL (male) or ≥ 9.5 gm/dL (female)
   * Platelets ≥ 75,000 /mm3
   * Serum alanine transaminase (SGPT/ALT) < 5 x upper limit of normal (ULN)
   * Serum aspartate transaminase (SGOT/AST) < 5 x ULN
   * Bilirubin (total) < 2.5 x ULN unless Gilbert's disease is present or subject is receiving atazanavir in the absence of other evidence of significant liver disease
   * Creatinine ≤ 1.5 x ULN
8. Clinically normal resting 12-lead ECG at Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator
9. Both male and female patients and their partners of childbearing potential must agree to use 2 medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], and intrauterine devices) during the course of the study (excluding women who are not of childbearing potential and men who have been sterilized). Females of childbearing potential must have a negative serum pregnancy test at Screening visit and negative urine pregnancy test prior to receiving the first dose of study drug.
10. Willing and able to participate in all aspects of the study, including use of SC medication, completion of subjective evaluations, attendance at scheduled clinic visits, and compliance with all protocol requirements as evidenced by providing written informed consent.

Note: Subjects diagnosed with either substance dependence or substance abuse or any history of a concomitant condition (e.g., medical, psychologic, or psychiatric) may be enrolled if in the opinion of site investigator these circumstances would not interfere with the subject's successful completion of the study requirements.

Exclusion Criteria:

1. Documented CXCR4-tropic virus or Dual/Mixed tropic (R5X4) virus
2. Patients with no viable treatment options (≤ 1 fully active drug)
3. Any active infection or malignancy requiring acute therapy (with the exception of local cutaneous Kaposi's sarcoma) Note: Subjects infected by the hepatitis B virus or early stage hepatitis C virus will be eligible for the study.
4. Laboratory test values of ≥ grade 3 DAIDS laboratory abnormality with the exception of the absolute CD4+ count criterion of < 200/mm3
5. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study
6. Unexplained fever or clinically significant illness within 1 week prior to the first study dose
7. Any vaccination within 2 weeks prior to the first study dose.
8. Subjects weighing < 35kg
9. History of anaphylaxis
10. History of Bleeding Disorder or patients on anti-coagulant therapy
11. Participation in an experimental drug trial(s) within 30 days of the Screening Visit or during the study
12. Any known allergy or antibodies to the study drug or excipients
13. Treatment with any of the following:

    * Radiation or cytotoxic chemotherapy with 30 days prior to the Screening Visit or during the study
    * Immunosuppressants within 60 days prior to the Screening Visit or during the study
    * Immunomodulating agents (e.g., interleukins, interferons), hydroxyurea, or foscarnet within 60 days prior to the Screening Visit or during the study
    * Oral or parenteral corticosteroids within 30 days prior to the Screening Visit or during the study. Subjects on chronic steroid therapy > 5 mg/day will be excluded with the following exception:

      * Subjects on inhaled, nasal, or topical steroids will not be excluded.
14. Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin DeJesus, MD, FACP,, Principal Investigator — Orlando Immunology Center
Locations (34):
- United States (32):
  - CD02 Investigational site, Fountain Valley, California
  - CD02 Investigational site, Long Beach, California
  - CD02 Investigational site, Los Angeles, California
  - CD02 Investigational Site, Los Angeles, California
  - CD02 Investigational site, Palm Springs, California
  - CD02 Investigational Site, San Francisco, California
  - CD02 Investigational site, San Francisco, California
  - CD02 Investigational Site, New Haven, Connecticut
  - CD02 Investigational site, Norwalk, Connecticut
  - CD02 Investigational Site, Washington D.C., District of Columbia
  - CD02 Investigational site, Washington D.C., District of Columbia
  - CD02 Investigational Site, Clearwater, Florida
  - CD02 Investigational site, Ft. Pierce, Florida
  - CD02 Investigational site, Miami, Florida
  - CD02 Investigational Site, Miami, Florida
  - CD02 Investigational site, Miami Beach, Florida
  - CD02 Investigational site, Orlando, Florida
  - CD02 Investigational site, West Palm Beach, Florida
  - CD02 Investigational site, Chicago, Illinois
  - CD02 Investigational site, Wichita, Kansas
  - E Study Site, Las Vegas, Nevada
  - CD02 Investigational site, New York, New York
  - CD02 Investigational site, Syracuse, New York
  - CD02 Investigational site, Charlotte, North Carolina
  - CD02 Investigational site, Cincinnati, Ohio
  - CD02 Investigational Site, Austin, Texas
  - CD02 Investigational Site, Bellaire, Texas
  - CD02 Investigational site, Dallas, Texas
  - CD02 Investigational Site, Houston, Texas
  - CD02 Investigational site, Houston, Texas
  - CD02 Investigational Site, Annandale, Virginia
  - CD02 Investigational Site, Spokane, Washington
- Puerto Rico (2):
  - CD02 Investigational site, Ponce, PR
  - CD02 Investigational site, San Juan

REFERENCES:
- [Derived] Gathe JC, Dejesus E, Ramgopal MN, Rolle CP, Yang OO, Sanchez WE, Lalezari JP, Krishen A, Sacha JB, Hansen SG, Meidling J. Leronlimab Treatment for Multidrug-Resistant HIV-1 (OPTIMIZE): A Randomized, Double-Blind, Placebo-Controlled Trial. J Acquir Immune Defic Syndr. 2025 Jun 1;99(2):185-194. doi: 10.1097/QAI.0000000000003648. PMID 39972543

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from U.S. sites only. The first participant was enrolled on 21 October 2015 and the last subject completed the study on 25 July 2018.
Pre-assignment Details: 365 participants were screened.
Groups:
- Placebo: Placebo weekly SC Inj. + existing ART for one week. After one week, all subjects will enter the 24-week single-arm, open-label treatment period. During this period, all subjects will receive PRO 140 SC injection and Optimized Background Therapy.
  Placebo
  Optimized Background Regimen: Optimized background therapy (OBT) is chosen on the basis of a subject's resistance test results and treatment history.
Period: Part 1 One-week Randomized
Arm/Group | PRO 140 | Placebo
Started | 25 | 27
Completed | 25 | 26
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Part 2 Open Label Treatment Period
Arm/Group | PRO 140 | Placebo
Started | 25 (In Open Label Treatment Period, all study participants received PRO140) | 26 (In Open Label Treatment Period, all study participants received PRO140)
Completed | 25 | 21
Not Completed | 0 | 5
Not completed — Non-medical | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Subject non compliant | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat: The Intent-to-Treat (ITT) population was defined as the set of subjects who were randomized and had received at least one (1) dose of leronlimab (PRO 140) or placebo. This population was to be used as the primary analysis population for the primary and secondary endpoints
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO 140 | Placebo | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (8.6) | 52.4 (6.7) | 52.4 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 17 | 21 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 13 | 24
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 27 | 52
Time since HIV Diagnosis [Mean (Standard Deviation); unit: years] | 20.0 (9.5) | 20.8 (9.4) | 20.4 (9.4)
Lowest CD4+ Cell Count [Count of Participants; unit: Participants]
  <200 cells/mm^3 | 10 | 12 | 22
  200-500 cells/mm^3 | 13 | 14 | 27
  >500 cells/mm^3 | 2 | 1 | 3
Number of ART Drug Exposure Prior to Enrollment [Mean (Standard Deviation); unit: Number of ART Drugs prior to enrolment] | 11.8 (4.8) | 9.6 (4.2) | 10.7 (4.6)
Number of ART Drug with Documented Resistance [Mean (Standard Deviation); unit: Number of ART drugs with resistance] | 9.4 (5.8) | 8.8 (3.3) | 9.1 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With ≥ 0.5 log10 Reduction in HIV-1 RNA Viral Load From Baseline at the End of the 1-week Double-blind Treatment Period
Description: The primary efficacy endpoint will be proportion of participants with a 0.5 log10 or greater reduction in HIV-1 RNA viral load from baseline at the end of the one week double-blind treatment period (Part 1).
Time Frame: From baseline visit to week 1 visit
Population: The primary population used for this analysis was the ITT population, defined as subjects who were randomized and had received at least one (1) dose of leronlimab (PRO 140) or placebo
Measure: Number; unit: Proportion of subjects
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 25 | 27
Proportion of subjects
  With >= 0.5 LOG10 IN HIV-1 RNA VIRAL Load Change from Baseline | .64 | .23
  Without >= 0.5 LOG10 IN HIV-1 RNA VIRAL Load Change from Baseline | .36 | .77
Statistical Analysis 1: Comparison: PRO 140 vs Placebo; Test type: Superiority; p = .0032, Fisher Exact; The Fisher's Exact test if the count in any cell was less than 5; otherwise Chi-Square test was to be used

2. Secondary Outcome: Proportion of Participants With ≥ 0.5 log10 Reduction in HIV-1 RNA Viral Load From Baseline at the End of the 1-week Double-blind Treatment Period, Stratified to Each Group: Resistance to ART Drugs Within Two Drug Class With Limited Treatment Option.
Description: Proportion of participants with ≥ 0.5 log10 reduction in HIV-1 RNA viral load from baseline at the end of the 1-week double-blind treatment period, stratified to each group:
  a. resistance to ART drugs within two drug class with limited treatment option (N = 24).
  This outcome measures the proportion of participants that are classified as having a resistance to ART drugs within two drug classes and with limited treatment options with ≥ 0.5 log10 reduction in HIV-1 RNA viral load from baseline at the end of the 1-week double-blind treatment period .
  The total number of participants in the study ITT population, 52, is further stratified into two subgroups:
  1. Participants with resistance to ART Drugs Within Two Drug Class With Limited Treatment Option (N = 24)
  2. Participants with resistance to ART Drugs Within Three Drug Classes (N = 28)
  This measure includes only the 24 participants with Resistance to ART Drugs Within Two Drug Class With Limited Treatment Options
Time Frame: From baseline visit to week 1 visit
Population: The total number of participants in the study ITT population, 52, is further stratified into two subgroups as follows:
  1. Participants with Resistance to ART Drugs Within Two Drug Class With Limited Treatment Option (N = 24)
  2. Participants with resistance to ART Drugs Within Three Drug Classes (N = 28)
  This measure includes only the 24 participants with Resistance to ART Drugs Within Two Drug Class With Limited Treatment Option
Measure: Number; unit: Proportion of participants
Groups:
- PRO 140: PRO140 350mg weekly SC Inj. + existing ART for one week. After one week, all subjects will enter the 24-week single-arm, open-label treatment period. During this period, all subjects will receive PRO 140 SC injection and Optimized Background Therapy.
  PRO 140: PRO 140 is a humanized IgG4,κ monoclonal antibody (mAb) to the chemokine receptor CCR5.
  A) Resistance to ART drugs within two drug class with limited treatment option.
- Placebo: Placebo weekly SC Inj. + existing ART for one week. After one week, all subjects will enter the 24-week single-arm, open-label treatment period. During this period, all subjects will receive PRO 140 SC injection and Optimized Background Therapy.
  Placebo
  A) Resistance to ART drugs within two drug class with limited treatment option.
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 11 | 13
Proportion of participants | .7273 | .2308
Statistical Analysis 1: Comparison: PRO 140 vs Placebo; Test type: Superiority; p = .0377, Fisher Exact

3. Secondary Outcome: Proportion of Participants With ≥ 0.5 log10 Reduction in HIV-1 RNA Viral Load From Baseline at the End of the 1-week Double-blind Treatment Period, Stratified to Each Group: Resistance to ART Drugs Within Three Drug Classes
Description: Proportion of participants with ≥ 0.5 log10 reduction in HIV-1 RNA viral load from baseline at the end of the 1-week double-blind treatment period, stratified to each group:
  a. Resistance to ART drugs within three drug classes (N = 28)
  This outcome measures the proportion of participants that are classified as having a resistance to ART drugs within two drug classes and with limited treatment options with ≥ 0.5 log10 reduction in HIV-1 RNA viral load from baseline at the end of the 1-week double-blind treatment period .
  The total number of participants in the study ITT population, 52, is further stratified into two subgroups as follows:
  1. Participants with Resistance to ART Drugs Within Two Drug Class With Limited Treatment Option (N = 24)
  2. Participants with resistance to ART Drugs Within Three Drug Classes (N = 28)
  This measure includes only the 28 participants with resistance to ART drugs within three drug classes
Time Frame: From baseline visit to week 1 visit
Population: The total number of participants in the study ITT population, 52, is further stratified into two subgroups as follows:
  1. Participants with resistance to ART Drugs Within Two Drug Class With Limited Treatment Options (N = 24)
  2. Participants with resistance to ART Drugs Within Three Drug Classes (N = 28)
  This measure includes only the 28 participants with resistance to ART drugs within three drug classes
Measure: Number; unit: Proportion of participants
Groups:
- PRO 140: PRO140 350mg weekly SC Inj. + existing ART for one week. After one week, all subjects will enter the 24-week single-arm, open-label treatment period. During this period, all subjects will receive PRO 140 SC injection and Optimized Background Therapy.
  PRO 140: PRO 140 is a humanized IgG4,κ monoclonal antibody (mAb) to the chemokine receptor CCR5.
  A) Resistance to ART drugs within three drug classes
- Placebo: Placebo weekly SC Inj. + existing ART for one week. After one week, all subjects will enter the 24-week single-arm, open-label treatment period. During this period, all subjects will receive PRO 140 SC injection and Optimized Background Therapy.
  Placebo
  A) Resistance to ART drugs within three drug classes
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 14 | 14
Proportion of participants | .5714 | .2308
Statistical Analysis 1: Comparison: PRO 140 vs Placebo; Test type: Superiority; p = .1201, Fisher Exact

4. Secondary Outcome: Mean Change From Baseline in HIV-1 RNA Levels (log10 Copies/mL) at the End of the 1-week Double-blind Treatment Period for All Patients and Within Each Stratum
Description: The raw and change from baseline in HIV-1 RNA levels (log10 copies/mL) at the end of the 1-week double-blind treatment period was to be summarized by treatment group for the first week during the double-blind treatment phase. For change from baseline summaries, subjects with an undefined change from baseline, because of missing data, were to be excluded. The change from baseline in HIV-1 RNA levels was to be compared between the two (2) groups using Analysis of covariance (ANCOVA) with the stratification factor (i.e., Resistance to ART drugs at the time of randomization) included in the model.
Time Frame: From baseline visit to week 1 visit
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Log10 Copies/mL
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 25 | 27
Log10 Copies/mL | 0.6 (0.45) | 0.1 (0.51)
Statistical Analysis 1: Comparison: PRO 140 vs Placebo; Test type: Superiority; p = .0013, ANCOVA

5. Secondary Outcome: Percentage of Participants Achieving HIV-1 RNA < 400 Copies/mL at Week 25 for All Patients and Within Each Stratum
Description: The number and percentages of subjects achieving HIV-1 RNA < 400 copies/mL at Week 25, from the open label portion of the study, are presented
Time Frame: 25 weeks
Population: The Intent-to-Treat (ITT) population was defined as the set of subjects who were randomized and received at least one (1) dose of leronlimab (PRO 140) or placebo
Measure: Count of Participants; unit: Participants
Groups:
- Part 2 Open Label Portion: 24-week single-arm, open-label treatment period with all subjects receiving PRO 140 along with OBT
Arm/Group | Part 2 Open Label Portion
Number analyzed (Participants) | 52
Participants
  With HIV-1 RNA < 400 Copies/mL at Week 25 | 37
  Without HIV-1 RNA < 400 Copies/mL at Week 25 | 3
  Missing | 12

6. Secondary Outcome: Percentage and Number of Participants Achieving HIV-1 RNA < 50 Copies/mL at Week 25 for All Patients and Within Each Stratum
Description: The number and percentages of subjects achieving HIV-1 RNA < 50 copies/mL at Week 25 are presented. This is from the 24 week open label portion of the of the trial.
Time Frame: 25 weeks
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Open Label Portion
Number analyzed (Participants) | 52
Participants
  With HIV-1 RNA < 50 Copies/mL at Week 25 | 32
  Without HIV-1 RNA < 50 Copies/mL at Week 25 | 8
  Missing | 12

7. Secondary Outcome: Mean Change From Baseline in HIV-1 RNA Levels (log10 Copies/mL) at Week 25 for All Patients and Within Each Stratum
Description: The raw and change from baseline in HIV-1 RNA levels (log10 copies/mL) at Week 25 was to be summarized for each week during the treatment phase. For change from baseline summaries, subjects with an undefined change from baseline, because of missing data, were to be excluded.
Time Frame: 25 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Part 2 Open Label Portion
Number analyzed (Participants) | 52
Log10 copies/mL | 2.4 (1.42)

8. Secondary Outcome: Mean Change From Baseline in CD4 Cell Count at the End of the 1-week Double-blind Treatment Period for All Patients and Within Each Stratum
Description: The raw and change from baseline in CD4 cell count at the end of the 1-week double blind treatment period was to be summarized by treatment group for the first week during the double-blind treatment phase. For change from baseline summaries, subjects with an undefined change from baseline, because of missing data, were to be excluded.
Time Frame: From baseline visit to week 1 visit
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: CD4 Cell Count
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 25 | 27
CD4 Cell Count | 41.1 (154) | 25 (131)
Statistical Analysis 1: Comparison: PRO 140 vs Placebo; The raw and change from baseline in CD4 cell count at the end of the 1-week double blind treatment period was to be summarized by treatment group for the first week during the double-blind treatment phase. For change from baseline summaries, subjects with an undefined change from baseline, because of missing data, were to be excluded; Test type: Superiority; p = .7123, ANCOVA

9. Secondary Outcome: Mean Change From Baseline in CD4 Cell Count at Week 25 for All Patients and Within Each Stratum
Description: The raw and change from baseline in CD4 cell count at Week 25 was to be summarized for each week during the treatment phase. For change from baseline summaries, subjects with an undefined change from baseline, because of missing data, were to be excluded.
Time Frame: 25 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: CD4 Cell Count
Arm/Group | Part 2 Open Label Portion
Number analyzed (Participants) | 52
CD4 Cell Count | 85.9 (175.2)

10. Secondary Outcome: Proportion of Participants With ≥ 1 log10 Reduction in HIV-1 RNA Viral Load From Baseline at the End of the 1-week Double-blind Treatment Period for All Patients and Within Each Stratum
Description: The number and percentage of subjects with a ≥ 1log10 or greater reduction in HIV-1 RNA viral load from baseline was to be presented for the two (2) treatment groups. The analysis of change in viral load was done for subjects with ≥ 1.0 log10 reduction in HIV-1 RNA after the first week of treatment. The analysis is presented for the ITT population
Time Frame: From baseline visit to week 1 visit
Population: as for outcome 5
Measure: Number; unit: Proportion of participants
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 25 | 27
Proportion of participants | .2 | .0385
Statistical Analysis 1: Comparison: PRO 140 vs Placebo; Test type: Superiority; p = .0993, Fisher Exact

11. Other Pre Specified Outcome: Tolerability of Repeated Subcutaneous Administration of PRO 140 as Assessed by Study Participants (Using Visual Analogue Scale) and by Investigator-evaluation of Injection Site Reactions
Description: Assessments of subject-perceived injection site pain using the Pain Visual Analog Scale (VAS) were performed during each visit to the clinic for a study visit.
  Beginning at Treatment Visit 2 (T2), subjects were asked to mark the point that best represents the average pain intensity over the past week at the injection site on a horizontal line (100 mm in length) anchored by the following word descriptors at each end, "no pain" on the left side and "pain as bad as it could possibly be" on the right side of the line. The subject marks on the line or by pointing to a position on the line the point that they feel represents their perception of their pain state. The VAS score is determined by measuring in millimeters from the left-hand end of the line to the point that the patient marks
  The scale range is 0mm to 100 mm, with 0 mm = No Pain and 100 mm = Pain as bad as it could possibly be.
  In this measurement, a lower number corresponds to less perceived pain.
  T# = Visit Week#
Time Frame: 25 weeks
Population: Assessments of subject-perceived injection site pain using the Pain Visual Analog Scale (VAS) was performed during each visit to the clinic for a study visit. The number of study participant visits varied each week and N = the number that visited the clinic and were assessed each week.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part 2 Open Label Portion
Number analyzed (Participants) | 50
Units on a scale
  T2 (Week 2) Left Side Injection Site | 1.3 (8.5)
  T2 (Week 2) Right Side Injection Site | 1.0 (7.1)
  T3 (Week 3) Left Side Injection Site: number analyzed (Participants) | 49
  T3 (Week 3) Left Side Injection Site | 0.3 (1.5)
  T3 (Week 3) Right Side Injection Site: number analyzed (Participants) | 49
  T3 (Week 3) Right Side Injection Site | 0.2 (0.7)
  T4 (Week 4) Left Side Injection Site: number analyzed (Participants) | 48
  T4 (Week 4) Left Side Injection Site | 0.4 (1.7)
  T4 (Week 4) Right Side Injection Site: number analyzed (Participants) | 48
  T4 (Week 4) Right Side Injection Site | 0.3 (1.1)
  T5 (Week 5) Left Side Injection Site: number analyzed (Participants) | 47
  T5 (Week 5) Left Side Injection Site | .7 (4)
  T5 (Week 5) Right Side Injection Site: number analyzed (Participants) | 47
  T5 (Week 5) Right Side Injection Site | .1 (.6)
  T6 (Week 6) Left Side Injection Site: number analyzed (Participants) | 49
  T6 (Week 6) Left Side Injection Site | .8 (4.8)
  T6 (Week 6) Right Side Injection Site: number analyzed (Participants) | 49
  T6 (Week 6) Right Side Injection Site | .3 (1.7)
  T7 (Week 7) Left Side Injection Site: number analyzed (Participants) | 48
  T7 (Week 7) Left Side Injection Site | .2 (.9)
  T7 (Week 7) Right Side Injection Site: number analyzed (Participants) | 48
  T7 (Week 7) Right Side Injection Site | .3 (1.7)
  T8 (Week 8) Left Side Injection Site | .3 (1.3)
  T8 (Week 8) Right Side Injection Site | .4 (1.5)
  T9 (Week 9) Left Side Injection Site: number analyzed (Participants) | 48
  T9 (Week 9) Left Side Injection Site | .2 (.8)
  T9 (Week 9) Right Side Injection Site: number analyzed (Participants) | 48
  T9 (Week 9) Right Side Injection Site | .2 (.9)
  T10 (Week 10) Left Side Injection Site: number analyzed (Participants) | 48
  T10 (Week 10) Left Side Injection Site | .3 (1.1)
  T10 (Week 10) Right Side Injection Site: number analyzed (Participants) | 48
  T10 (Week 10) Right Side Injection Site | .3 (1.1)
  T11 (Week 11) Left Side Injection Site: number analyzed (Participants) | 49
  T11 (Week 11) Left Side Injection Site | .3 (1.1)
  T11 (Week 11) Right Side Injection Site: number analyzed (Participants) | 49
  T11 (Week 11) Right Side Injection Site | .2 (1)
  T12 (Week 12) Left Side Injection Site: number analyzed (Participants) | 47
  T12 (Week 12) Left Side Injection Site | .9 (3)
  T12 (Week 12) Right Side Injection Site: number analyzed (Participants) | 47
  T12 (Week 12) Right Side Injection Site | .8 (2.7)
  T13 (Week 13) Left Side Injection Site: number analyzed (Participants) | 47
  T13 (Week 13) Left Side Injection Site | .1 (.9)
  T13 (Week 13) Right Side Injection Site: number analyzed (Participants) | 47
  T13 (Week 13) Right Side Injection Site | .1 (.9)
  T14 (Week 14) Left Side Injection Site: number analyzed (Participants) | 48
  T14 (Week 14) Left Side Injection Site | .4 (1.7)
  T14 (Week 14) Right Side Injection Site: number analyzed (Participants) | 48
  T14 (Week 14) Right Side Injection Site | .4 (1.8)
  T15 (Week 15) Left Side Injection Site: number analyzed (Participants) | 49
  T15 (Week 15) Left Side Injection Site | .1 (.6)
  T15 (Week 15) Right Side Injection Site: number analyzed (Participants) | 49
  T15 (Week 15) Right Side Injection Site | .2 (.9)
  T16 (Week 16) Left Side Injection Site: number analyzed (Participants) | 47
  T16 (Week 16) Left Side Injection Site | .4 (1.6)
  T16 (Week 16) Right Side Injection Site: number analyzed (Participants) | 47
  T16 (Week 16) Right Side Injection Site | .2 (.8)
  T17 (Week 17) Left Side Injection Site: number analyzed (Participants) | 45
  T17 (Week 17) Left Side Injection Site | .1 (.4)
  T17 (Week 17) Right Side Injection Site: number analyzed (Participants) | 45
  T17 (Week 17) Right Side Injection Site | .1 (.4)
  T18 (Week 18) Left Side Injection Site: number analyzed (Participants) | 46
  T18 (Week 18) Left Side Injection Site | .2 (1.2)
  T18 (Week 18) Right Side Injection Site: number analyzed (Participants) | 46
  T18 (Week 18) Right Side Injection Site | .3 (1.5)
  T19 (Week 19) Left Side Injection Site: number analyzed (Participants) | 48
  T19 (Week 19) Left Side Injection Site | .3 (1.3)
  T19 (Week 19) Right Side Injection Site: number analyzed (Participants) | 48
  T19 (Week 19) Right Side Injection Site | .2 (1.3)
  T20 (Week 20) Left Side Injection Site: number analyzed (Participants) | 45
  T20 (Week 20) Left Side Injection Site | 1.5 (8.9)
  T20 (Week 20) Right Side Injection Site: number analyzed (Participants) | 45
  T20 (Week 20) Right Side Injection Site | 1.1 (6)
  T21 (Week 21) Left Side Injection Site: number analyzed (Participants) | 45
  T21 (Week 21) Left Side Injection Site | .8 (4.5)
  T21 (Week 21) Right Side Injection Site: number analyzed (Participants) | 45
  T21 (Week 21) Right Side Injection Site | .4 (1.8)
  T22 (Week 22) Left Side Injection Site: number analyzed (Participants) | 44
  T22 (Week 22) Left Side Injection Site | .2 (.9)
  T22 (Week 22) Right Side Injection Site: number analyzed (Participants) | 44
  T22 (Week 22) Right Side Injection Site | .2 (.8)
  T23 (Week 23) Left Side Injection Site: number analyzed (Participants) | 46
  T23 (Week 23) Left Side Injection Site | .3 (1.7)
  T23 (Week 23) Right Side Injection Site: number analyzed (Participants) | 46
  T23 (Week 23) Right Side Injection Site | .2 (.9)
  T24 (Week 24) Left Side Injection Site: number analyzed (Participants) | 43
  T24 (Week 24) Left Side Injection Site | .2 (1.4)
  T24 (Week 24) Right Side Injection Site: number analyzed (Participants) | 43
  T24 (Week 24) Right Side Injection Site | 0 (.2)
  T25 (Week 25) Left Side Injection Site: number analyzed (Participants) | 44
  T25 (Week 25) Left Side Injection Site | .1 (.6)
  T25 (Week 25) Right Side Injection Site: number analyzed (Participants) | 44
  T25 (Week 25) Right Side Injection Site | 0 (.3)

12. Other Pre Specified Outcome: Frequency of Grade 3 or 4 Adverse Events as Defined by the DAIDS Adverse Event Scale
Description: The investigator was to carefully evaluate the comments of each subject and the response to treatment in order to judge the true nature and severity of the AE. The question of the relationship of AEs to study drug should have been determined by the investigator after thorough consideration of all available facts. To assess severity, the investigator was to use the DAIDS AE grading table for adverse events as well as any injection site reactions.
Time Frame: 25 weeks
Population: The Safety population was defined as all subjects who received at least one (1) dose of leronlimab (PRO 140) or placebo after randomization. This population was used for the analysis of safety parameters.
Measure: Number; unit: Number of Adverse Events
Arm/Group | Part 2 Open Label Portion
Number analyzed (Participants) | 52
Number of Adverse Events
  Moderate AEs | 40
  Severe AEs | 15

13. Other Pre Specified Outcome: Frequency of Treatment-Emergent Serious Adverse Events
Description: The incidence of serious adverse events (SAEs) by relationship to the study treatment. In total, there were 16 SAEs reported for eight (8) subjects (15.4%, 8/52). Thirteen of the SAEs were determined to be Unrelated, three were determined to be Unlikely Related to study treatment.
Time Frame: 25 weeks
Measure: Number; unit: Number of Serious Adverse Events
Arm/Group | Part 2 Open Label Portion
Number analyzed (Participants) | 52
Number of Serious Adverse Events
  Unrelated | 13
  Unlikely Related | 3

14. Other Pre Specified Outcome: Emergence of Dual/Mixed (D/M)- and CXCR4-tropic Virus in Patients Who Had Exclusive CCR5-tropic Virus at Study Entry.
Description: The number of study participants who had exclusive CCR5-tropic virus at study entry and subsequently developed Dual/Mixed (D/M)- and CXCR4-tropic virus at any time during study treatment while receiving PRO 140.
Time Frame: 25 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Open Label Portion
Number analyzed (Participants) | 52
Participants | 2

ADVERSE EVENTS:
Time Frame: 25 weeks
Description: Adverse events were systematically assessed through documented symptom-directed physical examinations, vital sign evaluation and injection site reaction evaluations performed at treatment and follow-up visits. All information is collected on case report forms.
Groups:
- Pro 140 Weekly for 1 Week; Part 2 PRO 140 Open Label for 24 Weeks: PRO140 350mg weekly SC Inj. + existing ART for one week. After one week, all subjects will enter the 24-week single-arm, open-label treatment period. During this period, all subjects will receive PRO 140 SC injection and Optimized Background Therapy.
  PRO 140: PRO 140 is a humanized IgG4,κ monoclonal antibody (mAb) to the chemokine receptor CCR5.
  Optimized Background Regimen: Optimized background therapy (OBT) is chosen on the basis of a subject's resistance test results and treatment history.
- Placebo Weekly for 1 Week: PRO140 350mg weekly SC Inj. + existing ART for one week. After one week, all subjects will enter the 24-week single-arm, open-label treatment period. During this period, all subjects will receive PRO 140 SC injection and Optimized Background Therapy.
  Placebo
  Optimized Background Regimen: Optimized background therapy (OBT) is chosen on the basis of a subject's resistance test results and treatment history.
Arm/Group | Pro 140 Weekly for 1 Week | Placebo Weekly for 1 Week | Part 2 PRO 140 Open Label for 24 Weeks
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27 | 8/52
Other Adverse Events (participants affected / at risk) | 2/25 | 2/27 | 34/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pro 140 Weekly for 1 Week (N=25) | Placebo Weekly for 1 Week (N=27) | Part 2 PRO 140 Open Label for 24 Weeks (N=52)
Pneumonia (Infections and infestations) | 0 | 0 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1
Schizoaffective disorder (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pro 140 Weekly for 1 Week (N=25) | Placebo Weekly for 1 Week (N=27) | Part 2 PRO 140 Open Label for 24 Weeks (N=52)
Fatigue (General disorders) | 1 | 0 | 3
Injection site haemorrhage (General disorders) | 0 | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Injection site pain (General disorders) | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Injection site bruising (General disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 2
Acute sinusitis (Infections and infestations) | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Hypotension (Vascular disorders) | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT02483078/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT02483078/SAP_001.pdf